CLINICAL TRIAL: NCT00710294
Title: DEBuT - HET: Device Based Therapy in Hypertension Extension Trial: Long-Term Follow-Up Trial for Patients Who Completed the DEBuT-HT Study
Brief Title: Device Based Therapy in Hypertension Extension Trial
Acronym: DEBuT-HET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360007-001
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension
Keywords: Refractory Hypertension; High Blood Pressure; Uncontrolled Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CVRx Rheos Baroreflex Hypertension Therapy System — The pulse generator, which is similar to a pacemaker, is typically implanted under the skin below the collarbone.
  Two small leads from the device are wrapped around the carotid arteries on both sides of the neck and connected to the pulse generator.
  Other Names: Rheos Hypertension Therapy; Baroreflex Activation Therapy™ (BAT™); Baroreflex Hypertension Therapy

SUMMARY:
This clinical investigation is designed to describe the long-term safety and efficacy of the CVRx Rheos Baroreflex Hypertension Therapy System in patients who participated in the DEBuT-HT study beyond the original follow up period (4-months or longer). The information obtained in this trial is intended to support regulatory approvals and market release of this therapy.

DETAILED DESCRIPTION:
This extension study, designed as a long-term follow up, will monitor the course of the disease and its treatment safety and efficacy by collecting the appropriate data and using data collected under the long term provisions of the DEBuT-HT study to describe and analyze the changes in ongoing drug treatment, the programming parameters of the implanted active device and any occurring adverse events over a period of up to 13 months after implant surgery in the DEBuT-HT trial. Annual follow-ups of up to five years are planned subsequently to the 13-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the follow-up period (4-month or longer) of the DEBuT-HT trial (protocol No.: 360004-001)
* Have signed an approved informed consent form for participation in this study

Exclusion Criteria:

* Are unable to comply with protocol requirements.
* Are enrolled in another concurrent clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Describe the safety of Rheos Baroreflex Hypertension Therapy System by evaluating all adverse events and estimating the system and procedure related adverse event rate until and including the 13-month follow-up. | after last 13-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Myriah Elletson, Study Chair — CVRx, Inc.
Locations (5):
- Germany (3):
  - University Hospital Bad Oeynhausen, Bad Oeynhausen
  - Charité Campus Buch, Berlin
  - University Hospital Hannover, Hanover
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- See also: Related Info — http://www.cvrx.com